CLINICAL TRIAL: NCT01973218
Title: A Phase 3, Randomized, Observer-blind, Multicenter Study to Evaluate the Immunogenicity and Safety of Novartis rMenB+OMV NZ Vaccine in Healthy Subjects Aged 11 to 17 Years in Korea
Brief Title: Safety and Immunogenicity Study of Two Doses of Novartis Meningococcal Serogroup B Recombinant Vaccine in Adolescents Aged 11-17 Years.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V72_42; 20130090378 (Other: MFDS)
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Meningococcal Disease
Keywords: Meningitis, adolescents, Meningococcal B
MeSH Terms: conditions — Meningococcal Infections; Meningitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rMenB (Experimental): Subjects received two doses of rMenB+OMV NZ vaccine (at Day 1 and Day 31) in the study.
  Interventions: Biological: Meningococcal B Recombinant vaccine rMenB+OMV NZ
- Placebo/MenACWY (Active Comparator): Subjects received one dose of saline placebo (Day 1) and one dose of MenACWY-CRM vaccine (Day 31) in the study.
  Interventions: Biological: Placebo; Biological: Meningococcal ACWY-CRM conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal B Recombinant vaccine rMenB+OMV NZ — Subjects were randomized to one of two treatment groups to receive intramuscular (IM) vaccination with two doses of rMenV+OMV NZ vaccine (0.5 mL) in the non-dominant arm, one month apart. Subjects were followed for two months.
  Arms: rMenB
Biological: Placebo — Subjects were randomized to one of two treatment groups to receive intramuscular (IM) injection of saline solution followed by one dose of MenACWY-CRM vaccine (0.5 mL), one month apart. Subjects were followed for two months.
  Arms: Placebo/MenACWY
Biological: Meningococcal ACWY-CRM conjugate vaccine — Subjects were randomized to one of two treatment groups to receive intramuscular (IM) injection of saline solution followed by one dose of MenACWY-CRM vaccine (0.5 mL), one month apart. Subjects were followed for two months.
  Other Names: Meningococcal (groups A,C,W,and Y) oligosaccharide diphtheria CRM-197
  Arms: Placebo/MenACWY

SUMMARY:
The purpose of the study was to assess the immunogenicity and safety of two doses of Novartis Meningococcal B Recombinant (rMenB+OMV NZ) vaccine administered one month apart (0, 1 month schedule) in Korean adolescents aged between 11 to 17 years.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents 11-17 years of age inclusive who have given their written assent and whose parent or legal guardian has given written informed consent at the time of enrollment;
2. Available for all the visits scheduled in the study (i.e. not planning to leave the area before the end of the study period);
3. In good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator;
4. With a negative urine pregnancy test (for female subjects only).

Exclusion Criteria:

1. History of any meningococcal vaccine administration;
2. Current or previous, confirmed or suspected disease caused by N. meningitidis;
3. Household contact with and/or intimate exposure to an individual with any laboratory confirmed N. meningitidis infection within 60 days of enrollment;
4. Pregnancy or nursing (breastfeeding) mothers;
5. Female subjects who have not used or do not plan to use acceptable birth control measures, for the 2 months duration of the study;
6. Any serious chronic or progressive disease;
7. Family members and household members of research staff;
8. Any condition which in the opinion of the investigator may interfere with the evaluation of the study objectives;
9. Significant acute or chronic infection within the previous 7 days or fever within 3 days prior to enrolment;
10. Antibiotics within 6 days prior to enrollment;
11. Known or suspected impairment/alteration of the immune system, immunosuppressive therapy;
12. Receipt of blood, blood products and/or plasma derivatives, or a parenteral immunoglobulin preparation within the previous 90 days;
13. History of severe allergic reactions after previous vaccinations or hypersensitivity to any vaccine component;
14. Receipt of or intent to immunize with any other vaccine(s) within 30 days prior and throughout the study period;
15. Participation in another clinical trial within the last 90 days or planned for during study.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 264 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (7):
- South Korea (7):
  - 06 Kosin University Gospel Hospital 34, amnam-dong, Seo-gu, Busan
  - 05 YuKorea University Ansan Hospital 23, Jeokgeum-ro, Danwon-gu, Ansan-si, Gyeonggi-do
  - 04 Pusan National University Yangsan Hospital 20 Geumo-ro, Mulgeum-eup, Yangsan, Gyeongsangnam-do
  - 07 Seoul National University Bundang Hospital 82, Gumi-ro 173 Beon-gil, Bundang-gu, Seongnam
  - 01 Seoul National University Hospital 101 Daehang-ro,, Jongno-gu, Seoul
  - 03 Ewha Womans University Mokdong Hospital, Department of Pediatrics, 911-1 Mokdong, Yangch’ŏn-gu, Seoul
  - 02 Inha University Hospital 7-206, 3rd street, Shinheung-dong, Jung-gu, Incheon

REFERENCES:
- [Derived] Lee HJ, Choe YJ, Hong YJ, Kim KH, Park SE, Kim YK, Oh CE, Lee H, Song H, Bock H, Casula D, Bhusal C, Arora AK. Immunogenicity and safety of a multicomponent meningococcal serogroup B vaccine in healthy adolescents in Korea--A randomised trial. Vaccine. 2016 Feb 24;34(9):1180-6. doi: 10.1016/j.vaccine.2016.01.033. Epub 2016 Jan 28. PMID 26826544

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 7 study sites in Korea.
Pre-assignment Details: All enrolled subjects were included in the trial.
Period: Overall Study
Arm/Group | rMENB | Placebo/MenACWY
Started | 176 | 88
Completed | 174 | 88
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rMENB | Placebo/MenACWY | Total
Number analyzed (Participants) | 176 | 88 | 264
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.5 (1.8) | 13.4 (1.8) | 13.5 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 36 | 113
  Male | 99 | 52 | 151

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Serum Bactericidal Antibody (SBA) Titers ≥1:4 Against Neisseria Meningitidis Serogroup B by Vaccine Group.
Description: Percentage of subjects with SBA titers ≥1:4 against each of the three indicators strains H44/76, 5/99 and NZ98/254 of N. Meningitidis serogroup B, at one month after second vaccination, are reported for each group.
Time Frame: Day 1 and Day 61
Population: Analysis was done on the Full Analysis Set (FAS) i.e. all subjects who received at least one study vaccine and had immunogenicity data at relevant timepoints.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | rMenb | Placebo/MenACWY
Number analyzed (Participants) | 174 | 88
percentage of subjects
  H44/76 strain (Day 1) | 26 [20 to 33] | 24 [15 to 34]
  H44/76 strain (Day 61) | 98 [97 to 99] | 27 [18 to 38]
  5/99 strain (Day 1) | 12 [8 to 18] | 10 [5 to 19]
  5/99 strain (Day 61) | 97 [93 to 99] | 16 [9 to 25]
  NZ98/254 strain (Day 1) | 16 [10 to 22] | 15 [8 to 24]
  NZ98/254 strain (Day 61) | 97 [93 to 99] | 17 [10 to 27]

2. Secondary Outcome: The SBA Geometric Mean Titers (GMTs) Against N.Meningitidis Serogroup B, by Vaccine Group.
Description: The SBA antibody titers against each of the three indicator strains of N.Meningitidis serogroup B at one month after second vaccination are reported as GMTs, for each group.
Time Frame: Day 1 and Day 61
Population: Analysis was done on FAS population, i.e. all subjects who received at least one study vaccine and had immunogenicity data at relevant timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | rMENB | Placebo/MenACWY
Number analyzed (Participants) | 174 | 88
Titers
  H44/76 strain (Day 1) | 2.31 [1.94 to 2.74] | 2.18 [1.72 to 2.77]
  H44/76 strain (Day 61) | 91 [74 to 112] | 2.56 [1.91 to 3.43]
  5/99 strain (Day 1) | 1.5 [1.31 to 1.72] | 1.37 [1.16 to 1.61]
  5/99 strain (Day 61) | 351 [284 to 432] | 1.84 [1.34 to 2.52]
  NZ98/254 strain (Day 1) | 1.71 [1.45 to 2.02] | 1.59 [1.27 to 1.99]
  NZ98/254 strain (Day 61) | 32 [26 to 40] | 1.77 [1.35 to 2.32]

3. Secondary Outcome: The Geometric Mean Ratio (GMR) of Post- Versus Pre-vaccination SBA Titers Against N.Meningitidis Serogroup B, by Vaccine Group.
Description: The GMR of post-vaccination versus pre-vaccination SBA titers against each of the three indicator strains of N.Meningitidis serogroup B, at one month after second vaccination (day 61/day 1) are reported, for each group.
Time Frame: Day 61/ Day 1
Population: Analysis was done on the FAS population, i.e. all subjects who received at least one study vaccine and had immunogenicity data at relevant timepoints
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | rMENB | Placebo/MenACWY
Number analyzed (Participants) | 174 | 88
Ratio
  H44/76 strain | 40 [32 to 49] | 1.18 [0.92 to 1.51]
  5/99 strain | 234 [181 to 301] | 1.34 [1.0 to 1.81]
  NZ98/254 strain | 19 [15 to 23] | 1.11 [0.92 to 1.35]

4. Secondary Outcome: The Percentages of Subjects With a Four-fold Increase in SBA Antibody Titers Against N.Meningitidis Serogroup B, by Vaccine Group.
Description: Percentages of subjects with a four-fold increase in SBA antibody titers from baseline against each of the three indicator strains of N.Meningitidis serogroup B, at one month after second vaccination are reported, for each group.
Time Frame: Day 61
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | rMENB | Placebo/MenACWY
Number analyzed (Participants) | 174 | 88
percentage of subjects
  H44/76 strain | 93 [88 to 96] | 8 [3 to 16]
  5/99 strain | 97 [93 to 99] | 6 [2 to 13]
  NZ98/254 strain | 83 [76 to 88] | 6 [2 to 13]

5. Secondary Outcome: The ELISA Geometric Mean Concentrations (GMCs) Against Vaccine Antigen 287-953, by Vaccine Group.
Description: The GMCs against vaccine antigen 287-953 was measured by Enzyme-linked Immunosorbent Assay (ELISA) , at one month after second vaccination and are reported for each group.
Time Frame: Day 1 and Day 61
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | rMENB | Placebo/MenACWY
Number analyzed (Participants) | 172 | 88
IU/mL
  Day1 | 23 [22 to 24] | 26 [23 to 29]
  Day61 | 1208 [1025 to 1423] | 27 [23 to 32]

6. Secondary Outcome: The GMR of Post Versus Pre-vaccination ELISA GMCs Against Vaccine Antigen 287-953, by Vaccine Groups.
Description: The GMR of post versus pre-vaccination GMCs against vaccine antigen 287-953, measured by ELISA at one month after second vaccination (day 61/day 1) are reported for each group.
Time Frame: Day 61/Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | rMENB | Placebo/MenACWY
Number analyzed (Participants) | 172 | 88
Ratio | 52 [44 to 62] | 1.05 [0.9 to 1.22]

7. Secondary Outcome: The Number of Subjects Reporting Solicited Adverse Events After Each Study Vaccination, by Vaccine Group.
Description: The number of subjects reporting solicited local and systemic adverse events (AEs) following rMenB+OMV NZ vaccination or placebo/MenACWY-CRM, are reported.
Time Frame: Day 1 through day 7 after each vaccination
Population: Analysis was done on the safety set for solicited AEs i.e all subjects in the Exposed Set who received the correct vaccination and provide post vaccination reactogenicity data.
Measure: Number; unit: Number of subjects
Arm/Group | rMENB | Placebo/MenACWY
Number analyzed (Participants) | 174 | 88
Number of subjects
  Any Local (1st vacc; N=174, 87) | 160 | 22
  Injec site pain (1st vacc; N=174,87) | 158 | 18
  Injec site erythema I (1st vacc; N=174,87) | 62 | 5
  Injec site erythema II (1st vacc; N=174,87) | 14 | 0
  Injec site swelling I (1st vacc; N=174,87) | 57 | 0
  Injec site swelling II (1st vacc; N=174,87) | 19 | 0
  Injec site induration I (1st vacc; N=174,87) | 55 | 3
  Injec site induration II (1st vacc; N=174,87) | 29 | 0
  Any Local (2nd vacc; N=173,88) | 145 | 36
  Injec site pain (2nd vacc; N=173,88) | 142 | 33
  Injec site erythema I (2nd vacc; N=173,88) | 49 | 17
  Injec site erythema II (2nd vacc; N=173,88) | 11 | 7
  Injec site swelling I (2nd vacc; N=173,88) | 47 | 16
  Injec site swelling II (2nd vacc; N=173,88) | 16 | 3
  Injec site induration I (2nd vacc; N=172,88) | 54 | 17
  Injec site induration II (2nd vacc; N=172,88) | 26 | 7
  Any Systemic (1st vacc; N=174,87) | 89 | 31
  Loss of appetite (1st vacc; N=174,87) | 15 | 8
  Nausea (1st vacc; N=174,88) | 20 | 7
  Malaise (1st vacc; N=174,87) | 51 | 13
  Myalgia (1st vacc; N=174,87) | 45 | 10
  Arthralgia (1st vacc; N=174,87) | 14 | 4
  Headache (1st vacc; N=174,87) | 42 | 19
  Body Temperature (≥38°C) (1st vacc; N=174,87) | 6 | 1
  Prevention of pain/fever (1st vacc;N=174,87) | 1 | 0
  Treatment of pain/fever (1st vacc;N=174,87) | 11 | 1
  Medically attended fever (1st vacc;N=174,86) | 1 | 0
  Any Systemic (2nd vacc; N=173,88) | 74 | 21
  Loss of appetite (2nd vacc; N=173,88) | 21 | 4
  Nausea (2nd vacc; N=173,88) | 15 | 5
  Malaise (2nd vacc; N=173,88) | 47 | 10
  Myalgia (2nd vacc; N=173,88) | 29 | 9
  Arthralgia (2nd vacc; N=173,88) | 15 | 7
  Headache (2nd vacc; N=173,88) | 50 | 16
  Body Temperature (≥38°C) (2nd vacc; N=173,88) | 9 | 1
  Prevention of pain/fever (2nd vacc;N=173,88) | 1 | 0
  Treatment of pain/fever (2nd vacc;N=173,88) | 12 | 1
  Medically attended fever (2nd vacc;N=171,88) | 2 | 0

8. Secondary Outcome: The Number of Subjects Reporting Unsolicited AEs After Any Vaccination, by Vaccine Group.
Description: The number of subjects reporting any unsolicited AEs, serious adverse events (SAEs), AEs leading to premature withdrawal and medically attended AEs (throughout the study), following rMenB+OMV NZ vaccination or placebo/MenACWY-CRM, are reported.
Time Frame: Day 1 through Day 61
Population: as for outcome 7
Measure: Number; unit: number of subjects
Arm/Group | rMENB | Placebo/MenACWY
Number analyzed (Participants) | 174 | 88
number of subjects
  Any AE | 45 | 10
  Possibly or Probably Related AES | 30 | 3
  SAEs | 2 | 0
  At least possibly related SAEs | 0 | 0
  Deaths | 0 | 0
  Medically attended AEs | 45 | 20
  AEs resulting in premature withdrawal | 1 | 0

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected between Day 1 to 7 after each vaccination; any unsolicited AEs (including serious AEs, medically attended AEs and AE's leading to premature withdrawal) from Day 1 to Day 61 (throughout the study)
Groups:
- Total: Total of subjects
Arm/Group | rMENB | Placebo/MenACWY | Total
Serious Adverse Events (participants affected / at risk) | 2/174 | 0/88 | 2/262
Other Adverse Events (participants affected / at risk) | 167/175 | 63/88 | 230/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rMENB (N=174) | Placebo/MenACWY (N=88) | Total (N=262)
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 1
PAROVARIAN CYST (Reproductive system and breast disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rMENB (N=175) | Placebo/MenACWY (N=88) | Total (N=263)
NAUSEA (Gastrointestinal disorders) | 30 | 10 | 40
INJECTION SITE ERYTHEMA (General disorders) | 25 | 8 | 33
INJECTION SITE INDURATION (General disorders) | 43 | 7 | 50
INJECTION SITE PAIN (General disorders) | 166 | 48 | 214
INJECTION SITE SWELLING (General disorders) | 31 | 4 | 35
MALAISE (General disorders) | 77 | 17 | 94
PYREXIA (General disorders) | 16 | 2 | 18
NASOPHARYNGITIS (Infections and infestations) | 16 | 14 | 30
EATING DISORDERS (Psychiatric disorders) | 29 | 11 | 40
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 26 | 11 | 37
MYALGIA (Musculoskeletal and connective tissue disorders) | 60 | 15 | 75
HEADACHE (Nervous system disorders) | 78 | 31 | 109

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial.